CLINICAL TRIAL: NCT01547767
Title: Investigations Into ISCU Myopathy or Iron Sulfur Scaffold U Protein Myopathy
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120062; 12-CH-0062
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Myopathy
Keywords: Metabolism; Muscle; Mutation; ISCU Myopathy; Myopathy
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other

SUMMARY:
Background:

- A mutation in a gene known as ISCU was found to be the cause of a rare myopathy that affects the muscles. Researchers collected clinical samples from people with this myopathy. More research is being done to develop a therapy for this disease. Researchers are asking for permission to study the samples already collected.

Objectives:

- To allow researchers to use clinical samples collected to study new treatments for ISCU myopathy.

Eligibility:

- People with ISCU myopathy who have provided clinical samples for study.

Design:

* Participants will allow researchers to study clinical samples already collected. Blood, urine, muscle, and cell samples may be used. Medical records and photographs may also be studied.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
In 2008, NIH investigators collaborated to find a mutation in the human gene, ISCU, which is the official human gene name for a gene involved in assembly of iron sulfur clusters, and is abbreviated from Iron Sulfur Cluster assembly protein, U, which was identified as the cause of a rare myopathy that affected about 25 patients in Sweden. This protocol is intended to allow for the collection and analysis of clinical specimens and medical information from several research subjects who previously participated in studies that led to identification of the disease gene.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects will be eligible for this study if they have ISCU myopathy or carry a mutation in ISCU.

No exclusions will be made based on gender or, ethnicity and adults

will be the only patients included.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey A Rouault, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Mochel F, Knight MA, Tong WH, Hernandez D, Ayyad K, Taivassalo T, Andersen PM, Singleton A, Rouault TA, Fischbeck KH, Haller RG. Splice mutation in the iron-sulfur cluster scaffold protein ISCU causes myopathy with exercise intolerance. Am J Hum Genet. 2008 Mar;82(3):652-60. doi: 10.1016/j.ajhg.2007.12.012. Epub 2008 Feb 14. PMID 18304497
- [Background] LARSSON LE, LINDERHOLM H, MUELLER R, RINGQVIST T, SOERNAES R. HEREDITARY METABOLIC MYOPATHY WITH PAROXYSMAL MYOGLOBINURIA DUE TO ABNORMAL GLYCOLYSIS. J Neurol Neurosurg Psychiatry. 1964 Oct;27(5):361-80. doi: 10.1136/jnnp.27.5.361. No abstract available. PMID 14213465
- [Background] Haller RG, Henriksson KG, Jorfeldt L, Hultman E, Wibom R, Sahlin K, Areskog NH, Gunder M, Ayyad K, Blomqvist CG, et al. Deficiency of skeletal muscle succinate dehydrogenase and aconitase. Pathophysiology of exercise in a novel human muscle oxidative defect. J Clin Invest. 1991 Oct;88(4):1197-206. doi: 10.1172/JCI115422. PMID 1918374
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-CH-0062.html